CLINICAL TRIAL: NCT01155063
Title: A Non-Interventional Observational Study Evaluating The Effects Of Exemestane Following 2-3 Years Of Adjuvant Tamoxifen Therapy On Safety In Postmenopausal And Hormone Receptors Positive Early Breast Cancer Patients
Brief Title: Evaluating The Safety Of Exemestane Following 2-3 Years Of Adjuvant Tamoxifen Therapy In Postmenopausal Early Breast Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5991092
Record Dates: First submitted 2010-06-28; First posted 2010-07-01 (Estimated); Results first posted 2012-09-20 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Early Breast Cancer
Keywords: Exemestane; Adjuvant Treatment In Postmenopausal Women; Estrogen Receptor Positive Early Breast Cancer; Tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Main Group: Postmenopausal Women With Invasive, Estrogen Receptor Positive Early Breast Cancer Who Are Disease-Free After 2-3 Years Of Initial Adjuvant Tamoxifen Therapy
  Interventions: Other: Aromasin (exemestane)

INTERVENTIONS:
Other: Aromasin (exemestane) — Aromasin (exemestane), tablets 25 mg, once a day
  Other Names: Aromasin, exemestane

SUMMARY:
Evaluating the safety, tolerability and efficacy of Aromasin® when used in routine clinical practice, evaluating adherence to prescribed Aromasin® treatment and to understand reasons for early discontinuation.

DETAILED DESCRIPTION:
This study was terminated on 01-Aug-2011 due to very low potential to enroll planned number of patients or any sufficient number of patients for complete statistical analyses. This study is not being terminated because of safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females.
* Patients who have had surgical treatment for histological confirmed breast cancer that was non-metastatic at the time of the initial diagnosis.
* Patients who are disease-free after 2 or 3 years of adjuvant tamoxifen treatment.
* Patients whose tumour was estrogen receptor positive (ER+).
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients for whom Aromasin® treatment is contraindicated (see SPC).
* Presence of metastasis or a contra lateral tumour.
* Other adjuvant endocrine therapy.
* Another concomitant antineoplastic treatment.
* Participation in a clinical trial with an investigational drug during the 30 days prior to enrolment in the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Postmenopausal Women With Invasive, Estrogen Receptor Positive Early Breast Cancer Who Are Disease-Free After 2-3 Years Of Initial Adjuvant Tamoxifen Therapy
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5991092&StudyName=Evaluating%20The%20Safety%20Of%20Exemestane%20Following%202-3%20Years%20Of%20Adjuvant%20Tamoxifen%20Therapy%20In%20Postmenopausal%20Early%20Breast%20Cancer%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane: Participants with 2-3 years of initial adjuvant tamoxifen therapy who received exemestane (Aromasin) 25 milligram (mg) oral tablet once daily to complete 5 years of adjuvant hormonal therapy.
Period: Overall Study
Arm/Group | Exemestane
Started | 89
Completed | 0
Not Completed | 89
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Study terminated by sponsor | 87

BASELINE CHARACTERISTICS:
Groups:
- Exemestane: Participants with 2-3 years of initial adjuvant tamoxifen therapy who received exemestane (Aromasin) 25 mg oral tablet once daily to complete 5 years of adjuvant hormonal therapy.
Arm/Group | Exemestane
Number analyzed (Participants) | 89
Age Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 0
Type of Tumor [Number; unit: Participants] — Number of participants with different types of tumor such as; ductal carcinoma, lobular carcinoma, invasive ductal carcinoma, invasive lobular carcinoma, papillary carcinoma, medullary carcinoma, mucinous (colloid) carcinoma and others.
  Participants
    Ductal carcinoma | 5
    Lobular carcinoma | 6
    Invasive ductal carcinoma | 50
    Invasive lobular carcinoma | 20
    Papillary carcinoma | 0
    Medullary carcinoma | 5
    Mucinous (colloid) carcinoma | 2
    Other | 1
Type of Surgery [Number; unit: Participants] — Number of participants who had undergone different type of surgeries which included mammectomy, radical resection, radical mastectomy, mastectomy, mammectomy with lymphadenectomy, ovariectomy, mammectomy with lymph node dissection, mastectomy type madden of mammary gland.
  Participants | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Hormone Receptor Status [Number; unit: Participants] — Number of participants with positive or negative estrogen and progesterone receptors.
  Participants
    Estrogen receptor: Positive | 87
    Estrogen receptor: Negative | 1
    Estrogen receptor: Unknown | 1
    Progesterone receptor: Positive | 84
    Progesterone receptor: Negative | 4
    Progesterone receptor: Unknown | 1
Lymph Node Status [Number; unit: Participants] | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Tumor Node Metastasis (TNM) Stage [Number; unit: Participants] — TNM was based on size of tumor, if cancer cells had spread to nearby lymph nodes (LN), or distant (to other parts of the body) metastasis had occurred. Stages included: stage 0(no evidence of cancer cells), stage 1(T1N0M0), stage IIA(T0N1M0, T1N1M0, T2N0M0), stage IIB(T2N1M0, T3N0M0), stage IIIA(T0N2M0, T1N2M0, T2N3M0, T3N1orN2M0), stage IIIC(any TN3M0), stage IV(anyT anyNM1), where T0=early form of tumor, T1= <2 centimeter(cm), T2=2-5 cm, T3= >2 cm, T4=large sized tumor, N0=not spread to LN, N1=spread to 1 to 3,N2=spread to 4 to 9,N3=spread >10 axillary LN, M0=no metastasis, M1= Metastasis.
  Participants
    Stage I | 20
    Stage IIA | 42
    Stage IIB | 13
    Stage IIIB | 8
    Stage IV | 0
    Stage IIIA | 4
    Stage IIIC | 2
Histopathological Grade [Number; unit: Participants] — The grade of a cancer depends on what the cells look like and the growth-rate. Lower grade indicates a slower-growing cancer and a higher grade indicates a faster-growing one. Grade 1 (resemble normal cells, not growing rapidly), grade 2 (grow faster than normal cells), grade 3 and 4 (abnormal cells, grow and spread aggressively).
  Participants
    Grade 1 | 16
    Grade 2 | 43
    Grade 3 | 5
    Grade 4 | 0
    Unknown | 25
Number of participants on chemotherapy [Number; unit: Participants] — Number of participants who received chemotherapy. Chemotherapeutic drugs included cyclophosphamide, doxorubicin, 5-fluorouracil, paclitaxel, epirubicin, fluorouracil.
  Participants | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Number of participants on radiotherapy [Number; unit: Participants] — Number of participants who received radiotherapy as measured in radiations per centigray (Rads/cGy).
  Participants | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Concomitant morbidities in the past [Number; unit: Participants] — Participants who had a concomitant morbidity in the past; participants with more than one concomitant co-morbidity were counted for each of the co-morbidity classes applicable.
  Participants
    Myocardial infarction | 2
    Thyroid disorder | 1
    Cholecystitis | 1
    Drug hypersensitivity | 1
    Lipid metabolism disorder | 1
    Rheumatic fever | 1
    Neoplasm malignant | 1
    Rectal cancer | 1
    Reproductive tract disorder | 19
    Hypertension | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study medication in a participant who received study medication.
Time Frame: Month 0 up to Month 36 or early withdrawal
Population: Safety analysis set included participants who received at least one dose of the study medication during the observation period.
Measure: Number; unit: Participants
Arm/Group | Exemestane
Number analyzed (Participants) | 89
Participants | 7

2. Secondary Outcome: Number of Participants With Concomitant Morbidities
Description: Participants who had a concomitant morbidity during the study for any period of time; participants with more than one concomitant morbidity were counted for each of the concomitant morbidity classes applicable.
Time Frame: Month 0 up to Month 36 or early withdrawal
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Exemestane
Number analyzed (Participants) | 89
Participants
  Coronary artery disease | 14
  Thyroid disorder | 6
  Cholecystitis chronic | 1
  Cholelithiasis | 1
  Diabetes mellitus | 8
  Lipid metabolism disorder | 10
  Osteoporosis | 1
  Reproductive tract disorder | 11
  Hypertension | 37
  Varicose vein | 1

3. Secondary Outcome: Number of Participants With Concomitant Medications
Description: Concomitant medication (any medication other than, and in addition to, the study medication) taken for any period of time during the study and was coded by World Health Organization (WHO) medical dictionary.
Time Frame: Month 0 up to Month 36 or early withdrawal
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Exemestane
Number analyzed (Participants) | 89
Participants
  Acetylsalicylic acid | 4
  Bisoprolol fumarate | 4
  Calcitonin, salmon | 1
  Calcium D3 "stada" | 2
  Captopril | 1
  Diltiazem | 1
  Durapatite | 1
  Enalapril | 9
  Glibenclamide | 2
  Indapamide | 5
  Inosine | 1
  Levothyroxine sodium | 1
  Loratadine | 1
  Metoprolol tartrate | 1
  Nifedipine | 2
  Penicillin not otherwise specified (NOS) | 1
  Pentaerithrityl tetranitrate | 2
  Suguan | 1
  Tyrosine | 1
  Vinpocetine | 1
  Zoledronic acid | 1

4. Secondary Outcome: Percentage of Participants Who Discontinued the Study Medication
Time Frame: Month 0 up to Month 36 or early withdrawal
Population: Data was not analyzed as the study was terminated due to insufficient number of participants enrolled in the study.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Reasons for Discontinuation From Study Treatment
Time Frame: Month 0 up to Month 36 or early withdrawal
Population: Data was not analyzed as the study was terminated due to insufficient number of participants enrolled in the study.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Discontinuation of Study Medication
Time Frame: Month 0 up to Month 36 or early withdrawal
Population: Data was not analyzed as the study was terminated due to insufficient number of participants enrolled in the study.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Participants With Recurrent Disease
Description: Percentage of participants with confirmed recurrent disease at the end of the study (recurrence was defined as loco-regional and/or contralateral and/or distance metastases).
Time Frame: Month 36 or early withdrawal
Population: Data was not analyzed as the study was terminated due to insufficient number of participants enrolled in the study.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Exemestane
Serious Adverse Events (participants affected / at risk) | 1/89
Other Adverse Events (participants affected / at risk) | 6/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=89)
Appendicitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=89)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Migraine (Nervous system disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was prematurely discontinued, therefore not all data was analyzed and only one outcome measure timeframe was presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.